CLINICAL TRIAL: NCT05866484
Title: Testicular Sperm Aspiration (TESA) vs. Microfluidic Sperm Separation (MSS) in Couples With High Sperm DNA Fragmentation Undergoing ICSI: Which Approach is Better
Brief Title: Testicular Sperm Aspiration (TESA) vs. Microfluidic Sperm Separation (MSS)
Acronym: TESA vs Zymot
Status: Completed | Type: Observational
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Other Study IDs: 3277
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Infertility, Male; Azoospermia; Reproductive Disorder
MeSH Terms: conditions — Infertility, Male; Azoospermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TESA-ICSI: Compare ICSI outcomes with high Sperm DNA fragmentation undergoing TESA (testicular sperm extraction)
- Zymot-ICSI: Compare ICSI outcomes with high Sperm DNA fragmentation using microfluidic sperm separation device (Zymot)

SUMMARY:
Normal embryonic development relies on the correct transmission of genetic information, and sperm DNA plays a crucial part in this process. Causes of poor sperm DNA integrity include unhealthy lifestyles such as smoking and exposure to gonadotoxins, as well as, obesity, varicoceles, infections, advanced paternal age and systemic disorders. An increase in DNA fragmentation in sperm has been linked to lower fertilisation rate, poorer quality embryos, lower pregnancy rate, and high miscarriages rate.

The best way for sperm selection and processing in assisted reproductive technologies (ART) should be noninvasive and cost-effective. It should also make it possible to identify high-quality spermatozoa and produce more favorable results in terms of pregnancy and live birth rates.7 Meanwhile, the microfluidic sperm separation technology is a less expensive and less invasive alternative. This method allows for the selection of motile sperm that have a normal morphology, low levels of reactive oxygen species (ROS), and low DFI

ELIGIBILITY:
Inclusion Criteria:

* Men with high DNA fragmentation (>20%) undergoing TESA-ICSI or Zymot-ICSI

Exclusion Criteria:

* Spouse with advanced maternal age (> 40 years)
* Egg donation cycle

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This retrospective study will compare and investigate ICSI outcomes in couples with high sperm DNA fragmentation using either testicular sperm (TESA) or microfluidic sperm separation device (Zymot)
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate | approximately 8 weeks
  Compare clinical pregnancy rate in couples with high Sperm DNA fragmentation

SECONDARY OUTCOMES:
Number of utilizable blastocysts obtained | Approximately 20 days
  Compare the number of utilizable embryos obtained in couples using TESA-ICSI vs Zymot-ICSI

CONTACTS AND LOCATIONS:
Overall Officials: Armand Zini, MD, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No